CLINICAL TRIAL: NCT04323995
Title: Effectiveness of Sprint Interval Training on Anthropometric Measures Among Obese and Overweight Young Adults: A Systematic Review
Brief Title: Efficacy of Sprint Interval Training on Anthropometric Measures
Status: Completed | Type: Observational
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Principal Investigator, Universiti Tunku Abdul Rahman
Other Study IDs: UMFB1002
Record Dates: First submitted 2019-11-03; First posted 2020-03-27 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sprint Interval Training — Sprint interval training of 2 weeks and more.

SUMMARY:
Due to the rising problem of overweight and obesity, many strategies are implemented to combat this issue and one of the most common ways is exercise training. Aerobic exercise is a popular and effective conservative strategy for weight and adiposity management and commonly used exercise protocols are moderate-intensity continuous training (MICT) and interval training (IT). MICT is typically defined as continuous effort that elicits 55%-70% of the maximal heart rate or promotes oxygen consumption equivalent to 40%-60% of the maximum oxygen intake. IT involves repeated exercise with periods of recovery, which includes high intensity interval training (HIIT) and Sprint interval training (SIT). HIIT is exercising at 80% to 100% of maximal heart rate while SIT involves "all-out" or "supramaximal" effort at the intensity of 100% of maximal oxygen uptake. Multiple systematic reviews on the effect of SIT on aerobic capacity or comparisons between other forms of exercise protocols to reduce body adiposity has been conducted, but so far no systematic review has been carried out to evaluate the efficacy of this protocol solely on anthropometric measures on young obese and overweight adults alone. Hence, in this study, a systematic review of the effect of SIT on anthropometric measurements in young obese or overweight adults will be reviewed, filtered and assembled.

DETAILED DESCRIPTION:
Keywords using "obese", "overweight", "sprint interval training", "interval training", "anthropometric measures","body mass index", "fat %" lean muscle mass will be searched through e-databases namely Pubmed (including MEDLINE), Pedro-search, Science Direct, Google Scholar, Web of Science, Scopus and Cochrane Library for the suitable original full text studies. Only randomized control trails will be included in this study and the "Tool for the assEssment of Study qualiTy and reporting in EXercise" (TESTEX) would be utilized to assess each individual study. TESTEX has been validated and is specific to exercise training. The authors wish to use TESTEX as it addresses several shortcomings that PEDro does not e.g. exercise adherence, withdrawal, relative exercise training intensity. In addition, study quality assessment of training studies is more robust with TESTEX. 2 independent evaluators will examine and screen each study for its efficacy to be included in the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals aged 18-35 years old
* Overweight individuals with a BMI of 25.0 to <30
* Obese individuals with a BMI of 30.0 or higher
* Original full texts with SIT as intervention, occurring 2 weeks or more

Exclusion Criteria:

* Male and female individuals aged below 18 and above 35 years old
* SIT as intervention, occurring less than 2 weeks

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Overweight and obese young adults, aged 18-35 years, who had participated in SIT training protocol for at-least 2 weeks or more. Changes in the anthropometric measures will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
BMI for change | At baseline (before intervention begin) and post training.
Fat % for change | At baseline (before intervention begin) and post training.
Lean Muscle Mass | At baseline (before intervention begin) and post training.
Waist Circumference for change | At baseline (before intervention begin) and post training.
Waist to hip ratio for change | At baseline (before intervention begin) and post training.

CONTACTS AND LOCATIONS:
Overall Officials: Imtiyaz Ali Mir, Principal Investigator — Universiti Tunku Abdul Rahman
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No